CLINICAL TRIAL: NCT00897871
Title: Pharmacokinetics and Pharmacogenetics of Anticancer Drugs in Infants and Young Children
Brief Title: Evaluating the Side Effects and How Well Anticancer Drugs Work in Very Young Patients With Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CCLG-PK-2006-09; CDR0000560121 (Registry Identifier: PDQ (Physician Data Query)); EU-20742; EUDRACT-2006-002845-36
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2009-06

CONDITIONS: Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific
MeSH Terms: interventions — Carboplatin; Cyclophosphamide; etoposide phosphate; Gene Expression Profiling; Amplified Fragment Length Polymorphism Analysis

INTERVENTIONS:
Drug: carboplatin
Drug: cyclophosphamide
Drug: etoposide phosphate
Genetic: gene expression analysis
Genetic: polymorphism analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Studying samples of blood in the laboratory from young patients with cancer may help doctors learn how carboplatin, cyclophosphamide, and etoposide affect the body and how patients will respond to treatment.

PURPOSE: This laboratory study is evaluating the side effects and how well anticancer drugs work in very young patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Investigate inter-individual variability in the pharmacokinetics of selected anticancer drugs in infants and children age < 2 years on current dosing schedules.
* Compare drug exposures and degree of pharmacokinetic variability in children < 2 years with data obtained from published studies in older children.
* Relate inter-individual variability in pharmacokinetics and drug exposure to clinical toxicity and response.
* Use pharmacokinetic data in conjunction with clinical information obtained following treatment to investigate the suitability of current dosing regimens in infants and young children.

OUTLINE: This is a multicenter study. Patients are stratified according to age in months (0 to 6 vs 6 to 12 vs 12 to 24).

Patients receive carboplatin, cyclophosphamide, or etoposide according to the dosing regimen detailed in the clinical protocol on which the child is being treated.

Blood samples are collected from patients receiving 1 of the 3 drugs by central venous catheter periodically during treatment to measure pharmacokinetics of the specific drug. Additional blood samples are collected for DNA extraction and polymorphism analysis in CYP2B6, CYP2C9, and other metabolizing enzymes in addition to the determination of the genetic variation in multiple drug resistance.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of childhood cancer
* Receiving carboplatin, cyclophosphamide, or etoposide as standard treatment as part of a clinical study at a Children's Cancer and Leukemia Group (CCLG) center

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Single or double lumen central venous catheter in place
* No concurrent anticonvulsants, azole antifungal agents, or chronic steroid treatment

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2007-02

PRIMARY OUTCOMES:
Pharmacokinetic parameters
Pharmacokinetic modelling comparing pharmacokinetic parameters to investigate the key factors involved in determining individual exposures to parent drugs and metabolites
Influence of pharmacokinetic parameters and genotype for metabolizing enzyme on event-free survival
Influence of pharmacokinetic parameters and genotype for metabolizing enzyme on toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Gareth Veal, Principal Investigator — University of Newcastle Upon-Tyne
Locations (21):
- Our Lady's Hospital for Sick Children Crumlin, Dublin, Ireland
- United Kingdom (20):
  - Birmingham Children's Hospital, Birmingham, England
  - Bristol Royal Hospital for Children, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - University College Hospital, London, England
  - Great Ormond Street Hospital for Children, London, England
  - Royal Manchester Children's Hospital, Manchester, England
  - Sir James Spence Institute of Child Health at Royal Victoria Infirmary, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales